CLINICAL TRIAL: NCT06967961
Title: Research of Double-positive Circulating Cells (Tumor Marker / CD45+) in Several Types of Metastatic Cancers
Acronym: DP-PAN-CANCER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24GENE19
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Urothelial Carcinoma; Renal Cancer; Prostate Adenocarcinoma; Adenocarcinoma of Endometrium; Cutaneous Melanoma; Soft Tissue Sarcoma (STS); Nonseminomatous Germ Cell Tumor; Seminomatous Germ Cell Tumor; Upper Aerodigestive Tract Carcinoma; Cervical Carcinoma
Keywords: metastatic cancers; Double Positive Circulating cells; liquid biopsy
MeSH Terms: conditions — Carcinoma, Transitional Cell; Kidney Neoplasms; Melanoma; Sarcoma; Nonseminomatous germ cell tumor; Uterine Cervical Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with metastatic cancer (Other): * Blood sample collection for circulating DP cell detection by flow cytometry and Cell Search analysis for the following patients:
    * Cohort 1 : urothelial carcinoma
    * Cohort 2 : renal carcinoma
    * Cohort 3 : prostate adenocarcinoma
    * Cohort 4 : upper aerodigestive tract carcinoma
    * Cohort 5 : cervical carcinoma
    * Cohort 6 : adenocarcinoma of endometrium
  * Blood sample collection for circulating DP cell detection by flow cytometry and Parsotix analysis for the following patients:
    * Cohort 7 : cutaneous melanoma
    * Cohort 8 : soft tissue sarcoma
    * Cohort 9 : seminomatous and nonseminomatous germ cell tumors
  Interventions: Other: For each enrolled patient, the sample described below will be collected as specific intervention intended for research purposes:

INTERVENTIONS:
Other: For each enrolled patient, the sample described below will be collected as specific intervention intended for research purposes: — A blood sample will be taken before initiation of the metastatic treatment line and will be analyzed by 2 distinct methods. The total blood volume withdrawn per patient is approximately 30mL.

SUMMARY:
A prospective, proof-of-concept pilot study in patients with metastatic cancers (9 types of cancers are studied) treated at the IUCT-O or possibly in other institutions. Eligible patients will be selected and informed of this study during a medical consultation for their cancer by medical oncologists. Then, with the patient's consent and before the start of anti-cancer treatment (whatever the line), a blood sample will be taken to detect DP-circulating cells by 2 different methods of analysis.

Each patient will participate in the study for one day. The methods of analysis will be: flow cytometry for all patients and either Parsotix® or CellSearch® depending on the type of cancer.

450 patients will be enrolled in total.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with one of the following cancer types: urothelial carcinoma, renal carcinoma, prostate adenocarcinoma, upper aerodigestive tract carcinoma, cervival carcinoma, adenocarcinoma of endometrium, cutaneous melanoma, soft tissue sarcoma, seminomatous and nonseminomatous germ cell tumors
* 2. Metastatic disease for which the treatment (whatever the line) has not been initiated yet
* 3. Age ≥ 18 years
* 4. Patient affiliated to a French Social Security scheme
* 5. Patient having signed his/her informed consent prior to inclusion in the study and prior to any specific procedure for the study.

Exclusion Criteria:

* 1. Patient with localized disease.
* 2. Pregnant or breast-feeding women.
* 3. Any psychological, family, geographical or sociological condition that prevents compliance with the medical monitoring and/or procedures set out in the study protocol.
* 4. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2029-07-23 (Estimated); Study Completion 2029-07-23 (Estimated)

PRIMARY OUTCOMES:
Rate of patients presenting blood circulating DP cells detected by at least one of the two tested techniques (Flow Cytometry/ CellSearch® or Parsortix® according to the type of tumor) | 1 year after the Last Patient Last Visit
  It is defined as the ratio of number of patients for whom DP cells were detected (by at least 1 of the 2 techniques) by the total number of patients.

SECONDARY OUTCOMES:
Rate of patients presenting blood circulating DP cells detected by each method of analysis (Flow Cytometry and CellSearch® or Parsortix® according to the tumor type) | 1 year after the Last Patient Last Visit
  It is defined as the ratio of the number of patients presenting DP cells (detected by the concerned technique) by the total number of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Oncopole Claudius Regaud, IUCT-O, Toulouse, France